CLINICAL TRIAL: NCT07063407
Title: A Phase I Clinical Study Evaluating Safety, Tolerability, Pharmacokinetics and Efficacy of Intravenous HS-20093 Combinations in Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Phase 1 Study of HS-20093 Combinations in Patients With Extensive Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hansoh Biomedical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Hansoh BioMedical R&D Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-108
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Extensive Stage Small Cell Lung Cancer (ES-SCLC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HS-20093 and Adebrelimab (Experimental)
  Interventions: Drug: HS-20093 in combination with Adebrelimab

INTERVENTIONS:
Drug: HS-20093 in combination with Adebrelimab — HS-20093 in combination with Adebrelimab will be administered intravenously every 3 weeks until disease progression or other criteria for termination of treatment are met.

SUMMARY:
This is a Phase I clinical study of HS-20093. The purpose of this study is to evaluate the safety, tolerability, PK and efficacy of HS-20093 in combination with Adebrelimab in patients with Extensive Stage Small Cell Lung Cancer (ES-SCLC).

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase I clinical study to evaluate the safety, tolerability, PK and efficacy of HS-20093 in combination with Adebrelimab in patients with ES-SCLC. Patients with ES-SCLC without disease progression after receiving first-line standard induction therapy (Platinum + Etoposide +PD- (L) 1 inhibitor combination therapy) will receive maintenance therapy of HS-20093 in combination with Adebrelimab. Patients will continue treatment until disease progression or other criteria for termination of treatment are met.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Men or women aged more than or equal to (≥) 18 years.
2. Pathologically diagnosed as ES-SCLC.
3. Without disease progression after receiving first-line standard induction therapy (Platinum + Etoposide +PD- (L) 1 inhibitor combination therapy).
4. Eastern Cooperative Oncology Group (ECOG) performance status: 0~1.
5. Estimated life expectancy >12 weeks.
6. Adequate bone marrow reserve or serious organ dysfunction
7. Reproductive-age women agree to use adequate contraception and cannot breastfeed while participating in this study and for a period of 6 months after the last dose. Likewise, men also consent to use adequate contraceptive method within the same time limit.
8. Females must have evidence of non-childbearing potential.
9. Signed and dated Informed Consent Form.

Exclusion Criteria:

1. Uncontrolled pleural effusion or ascites or pericardial effusion.
2. Known and untreated, or active central nervous system metastases.
3. Active autoimmune diseases or active infectious disease
4. Known to have interstitial pneumonia or immune pneumonia
5. History of severe allergic reaction, serious transfusion reactions or Allergy to any component of HS-20093
6. The subject who is unlikely to comply with study procedures, restrictions, or requirements judged by the investigator.
7. The subject whose safety cannot be ensured or study assessments would be interfered judged by the investigator.
8. Pregnant women, breastfeeding women or woman who has a child-bearing plan during the study.
9. History of neuropathy or mental disorders, including epilepsy and dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Pogression-free survival (PFS) determined by investigators according to RECIST 1.1 | up to approximately 24 months
  PFS is deﬁned as the time from date of ﬁrst dose until the documentation of objective PD or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From the first dose through 90 days post end of treatment
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered an investigational product, which may present with symptoms, signs, disease, or laboratory abnormalities, but do not necessarily have a causality with the investigational product.
Objective response rate (ORR) assessed by investigator | up to approximately 24 months
  ORR is defined as the percentage of patients with a CR or PR that is confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1
Disease Control Rate (DCR) | up to approximately 24 months.
  Disease control is deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 5 weeks).
Duration of response (DOR) | up to approximately 24 months.
  Duration of response assessed by RECIST 1.1. Duration of response is defined as the time from when the criteria for CR or PR were first met to the occurrence of an objective disease progression (PD) or death.
Overall survival (OS) | up to approximately 24 months.
  OS is defined as time from first study treatment to death due to any cause.
Observed maximum plasma concentration (Cmax) of HS-20093 | up to approximately 24 months.
  Cmax of HS-20093
Area Under the Plasma Concentration-Time Curve (AUC) of HS-20093 | up to approximately 24 months.
  AUC of HS-20093
Percentage of participants with antibodies to HS-20093 in serum | up to approximately 24 months.
  Serum samples were collected for the determination of anti-drug antibody (ADA) at designated time points

IPD SHARING:
Plan to Share IPD: Undecided